CLINICAL TRIAL: NCT04051177
Title: Theory-based HIV Disclosure Intervention for Parents
Acronym: ICOPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: Guangxi Zhuang Autonomous Region Center for Disease Prevention and Control (Other Government)
Responsible Party: Principal Investigator, Xiaoming Li, Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 10006371
Record Dates: First submitted 2019-04-10; First posted 2019-08-09 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-08

CONDITIONS: HIV/AIDS; Disclosure
Keywords: parental HIV disclosure; China; intervention
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- parents living with HIV intervention group (Experimental): Parents living with HIV in this group received five two-hour parent HIV disclosure intervention, delivered one session per week for five weeks in the clinics where the parents are recruited. The intervention curriculum is modeled after the TRACK program with supplemental materials from TALC.
  Interventions: Behavioral: Interactive Communication with Openness, Passion, and Empowerment "ICOPE"
- Parents living with HIV control group (Other): Parents living with HIV in this group received five two-hour nutrition education curriculum in same delivery way. The nutrition curriculum is modeled after the "Simply Good Eating: curriculum developed at University of Minnesota.
  Interventions: Behavioral: Nutrition Curriculum

INTERVENTIONS:
Behavioral: Interactive Communication with Openness, Passion, and Empowerment "ICOPE" — The parent curriculum consists of five interactive training sessions (120 minutes each session for 10 hours total) with three specific focuses: understanding the stages of childhood cognitive development in the context of parental illness (Session #1 "Child's readiness for disclosure"); improving the parents' cognitive and behavioral skills related to parental HIV disclosure (Session #2 "Benefits and risks of disclosure", Session #3 "How to tell and what to tell", and Session #4 "Disclosure is an ongoing process"); and improving parental psychosocial well-being in adapting to living with HIV/AIDS (Session #5 "Cope with my infection/illness"). The curriculum addresses the issues of child and family strengths and community support across sessions.
  Arms: parents living with HIV intervention group
Behavioral: Nutrition Curriculum — The modified curriculum consists of five 2-hour interactive training sessions with aims to increase parents' knowledge of nutrition (Session #1: Food variety; Session #2: Food for growing child), healthy diets and cooking practice (Session 3: Fat, salt and sugar; Session 4: Fruits, vegetables and minerals), and food safety (Session #5 "Food safety")
  Arms: Parents living with HIV control group

SUMMARY:
The investigators propose to develop, implement, and evaluate a theory-driven parental disclosure intervention to assist parents living with HIV (PLH) to make a planned, developmentally appropriate disclosure of their HIV status to their uninfected children or, for PLH with younger children, to articulate a clear plan for disclosure to their children when developmentally appropriate. The majority of the 33.4 million individuals living with HIV worldwide reside in low-resource settings and are also of reproductive and child-rearing age. It is therefore important to the field of public health to develop an evidence-based parental disclosure intervention that can be effectively delivered to parents by a broad range of paraprofessionals. The investigators hypothesize that the proposed intervention will demonstrate efficacy in helping PLH to make developmentally appropriate disclosure to children or make a developmentally appropriate plan of disclosure and will demonstrate short, medium, and long-term efficacy in improving the well-being of parents, children, and families. The proposed scientifically rigorous evaluation includes mixed methods of data collection, a cluster randomized controlled trial, multiple data sources, and a 36-month longitudinal follow-up involving a large sample of parents, children, and providers. The intervention program to be developed and the evaluation data to be collected in the current study will inform the practice and clinic guidelines aimed at improving both parental HIV disclosure and the well-being of PLH, children and families in China and other low-and middle-income countries (LMICs).

DETAILED DESCRIPTION:
Because programs preventing prenatal HIV transmission are reaching a greater number of pregnant women worldwide and are successfully reducing vertical transmission, an ever increasing majority of children born to HIV-positive mothers are uninfected. In addition, new medical innovations and increasing availability of antiretroviral therapy (ART) have improved the health and longevity of HIV-positive parents, which means they are more likely to raise their children for many years after the initial diagnosis. For parents living with HIV ("PLH"), disclosing their HIV infection to their seronegative children ("parental HIV disclosure") becomes an increasingly important issue in terms of well-being of parents, children and families. The global literature in parental HIV disclosure suggests that developmentally appropriate, well-planned disclosure can greatly benefit the well-being of PLH, their children and families. However, for multiple reasons including fear of stigma and the psychological burden such knowledge might place on their children, PLH often struggle about whether, when, what, and how to talk to their children about their HIV infection. Many of them do not disclose their HIV infection to children primarily because they lack the confidence and behavioral skills to appropriately and effectively accomplish this task. To date, the issues surrounding parental HIV disclosure have been understudied, particularly in low- and middle-income countries (LMICs) including China where the HIV epidemic has been steadily expanding. In this application, the investigators propose to adapt relevant components from two evidence-based programs developed in the US to produce a theory-driven developmentally appropriate parental HIV disclosure intervention in Guangxi, China, where the investigators have built a strong research infrastructure and community collaboration through NIH-funded research since 2004. The proposed project consists of three main operational phases. Phase I includes formative research to examine current practices, barriers and facilitators, cultural influences, and effects of disclosure on PLH and their children. The data to be collected in this phase will complement the data the investigators have collected and will inform the adaption of intervention content and delivery modality. Phase II includes the development and pilot-testing of a theory-guided parental HIV disclosure intervention program with two components (a primary parent component and a secondary care provider component) by culturally adapting and integrating aspects of two US-based programs that were efficacious in either helping parents to make appropriate HIV disclosure or improving mental health status of PLH and their children. Phase III will rigorously evaluate the efficacy of the proposed intervention on well-being of PLH, children and families over 36 months through a cluster randomized controlled trial involving 800 PLH (either fathers or mothers) and their children (6 to 15 years of age). The research will also identify contextual and individual factors that potentially mediate or moderate the effect of the proposed intervention on parent, child, and family outcomes. The proposed research will address the dearth of targeted interventions supporting parental efforts in disclosing their HIV status to their children by examining whether a theory-based intervention can improve parental HIV disclosure in a low-resource setting. The proposed study will also provide cross-cultural evidence to support the role of parental disclosure in the well-being of parents, children, and families.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age;
* a confirmed diagnosis of HIV or AIDS;
* living with at least one child 6 to 15 years of age;
* having not disclosed their HIV status to their children;
* willing to consent one child to participate in the study.

Exclusion Criteria:

* linguistic, mental or physical inability to respond to assessment questions or to participate in intervention;
* currently incarcerated or institutionalized for drug use or commercial sex;
* plan to permanently relocate outside of the province within a year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 791 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
number of participants who have disclosed their HIV serostatus to their children assessed by one question in the survey | from baseline to 36 month follow-up
  question in questionnaire "have you disclosed your HIV serostatus to your children"?
participants' stage status regarding parental disclosure assessed by one question in the survey with 6 stages (see description) | from baseline to 36 month follow-up
  question in questionnaire "what stage status are you in now regarding disclosing your status to your children" 1 = "having not started disclosure in the past 6 months and no intention to start", 2 = "having not started disclosure in the past 6 months but is intending to start", 3 = "having not started disclosure in the past 6 months but already made a plan", 4 = "started disclosing but not mentioning HIV", 5 = "started disclosing with the word HIV", and 6 = "started disclosing with the word HIV and how I got infected".

SECONDARY OUTCOMES:
depression | from baseline to 36 month follow-up
  The Center for Epidemiologic Studies Depression Scale. Depression is measured using the Center for Epidemiologic Studies Short Depression Scale (CES-D 10) with a 4-point ordinal response: 0 = rarely or none of the time (less than 1 day); 1 = some or a little of the time (1-2 days); 2 = occasionally or a moderate amount of the time (3-4 days); 3 = most or all of the time (5-7 days). A summary score of all 10 items is calculated with higher scores indicating higher levels of depression. The summary score ranges between 0 to 30, and a score of 10 or greater is considered depressed.
stress | from baseline to 36 month follow-up
  Perceived Stress Scale. Perceived stress is assessed using 14 items from the perceived stress scales (PSS) with a 5-point responses option (0 = never, 1 = almost never, 2 = sometimes, 3 = fairly often, 4 = very often). A composite score was calculated by summing all 14 item responses. The composite score ranges between 0 to 56, and Higher scores indicating a higher level of perceived stress.
tobacco use | from baseline to 36 month follow-up
  tobacco use
alcohol use | from baseline to 36 month follow-up
  alcohol use
drug use | from baseline to 36 month follow-up
  drug use
condom use in sexual intercourse | from baseline to 36 month follow-up
  condom use
quality of life of people living with HIV | from baseline to 36 month follow-up
  The Medical Outcomes Study HIV Health Survey is composed of 35 items with 3, 5, and 6-point likert-type scale and dichotomous yes/no. 11 of the 35 items in the survey require recoding. Item scores are linearly transformed to a 0-100 scale with higher score indicating a higher level of quality of life.
most recent CD4 count | from baseline to 36 month follow-up
  most recent CD4 count
most recent viral load | from baseline to 36 month follow-up
  most recent viral load
disease progression | from baseline to 36 month follow-up
  disease progression using the HIV staging system by WHO

CONTACTS AND LOCATIONS:
Locations (1):
- University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided